CLINICAL TRIAL: NCT00500240
Title: Effect of Tight Control of Blood Glucose During Hyper-CVAD Chemotherapy For Acute Lymphocytic Leukemia
Brief Title: Effect of Tight Control of Blood Glucose During Hyper-CVAD Chemotherapy For Acute Lymphocytic Leukemia (ALL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early due to futility.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0107
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia; Lymphoma
Keywords: Acute Lymphocytic Leukemia; Leukemia; Lymphoma; Burkitts Lymphoma; Lymphoblastic Leukemia; Blood Sugar; Hyperglycemia; Insulin Aspart; Insulin Glargine; Hyper-CVAD
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Hyperglycemia | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Care (No Intervention): Control Group: Conventional care using blood sugar management with regular human insulin.
- Intensive Insulin (Other): Intervention Group: Intense blood sugar management with Insulin Aspart + Insulin Glargine
  Interventions: Drug: Insulin Glargine; Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Glargine — Use of human insulin glargine for slow decrease of blood sugar level over 24 hours.
  Arms: Intensive Insulin
Drug: Insulin Aspart — Use of human insulin aspart for rapid lowering of the blood glucose level over 24 hours.
  Arms: Intensive Insulin

SUMMARY:
The goal of this clinical research study is to learn if intense management and control of blood sugar levels during treatment for acute lymphocytic leukemia, Burkitts lymphoma, or lymphoblastic lymphoma will result in decreased risk of relapse, fewer complications, and/or longer survival.

DETAILED DESCRIPTION:
High blood sugar is a common side effect of treatment for certain types of cancer.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive blood sugar management with regular human insulin. Participants in the other group will receive more intense management with two newer forms of human insulin - insulin aspart, for rapid lowering of the blood glucose and insulin glargine for the slow decrease of blood sugar level over 24 hours.

You will receive additional blood tests (about 1 tablespoon each) at the time of entry on the study and after about every 2 to 4 courses of chemotherapy while on the study. These blood tests help better define the severity of your high blood sugar and your body's ability to metabolize sugar. Any bone marrow and blood samples that were collected before your therapy for your leukemia may be used for lab tests to measure markers of glucose metabolism in the blood. You will not be required to have a bone marrow biopsy after enrollment on study.

While in the hospital receiving chemotherapy, you will have your blood sugar checked 3 to 4 times a day. To check your blood sugar level, you, your nurse, or a laboratory technician will prick your finger with a small needle and place a small drop of blood on a test strip. If your blood sugar is high, you will be given the appropriate amount of insulin.

Before you begin out-patient insulin treatment, a research nurse, doctor, or diabetes educator will watch how you and/or your caregiver administer your insulin shots, to make sure that it is done correctly and safely. Once you leave the hospital, you will be required to check your own blood sugar 3 times a day and take insulin (either yourself or with the help of a health provider) up to 4 times a day while on steroid therapy and for 2 days after receiving steroids. On all other days you will be required to check your blood glucose once or twice a day and administer insulin 1 - 3 times daily. You will also need to speak with a nurse by phone every 1-3 days for review of blood sugar measurements and possible adjustment of the dose of insulin you must take.

You will remain on the study from the time you are found to have high blood sugar levels until completion of your chemotherapy (about 8 months for most patients). You may be taken off this study at any time if you find that you are unable or unwilling to monitor your glucose or receive insulin shots at home.

You will be followed for high blood sugar levels while you are receiving treatment with Hyper-CVAD chemotherapy regimen (fractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating cycles with methotrexate, cytarabine, methylprednisolone). If you continue to have high blood sugar after completion of this treatment, you will have continued follow-up either with your primary physician at home or if you choose, in the Internal Medicine Clinic at M. D. Anderson.

This is an investigational study. All of the insulin used in this study is FDA approved for the treatment of high blood sugar and commercially available. A total of up to 114 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 15 years.
2. Previously untreated ALL, Burkitt's lymphoma, or lymphoblastic leukemia receiving induction chemotherapy with hyper-CVAD or variants of the hyper-CVAD regimen.
3. Random serum glucose >/= 180 mg/dL detected during the first 2 cycles of chemotherapy and confirmed with a second measurement.

Exclusion Criteria:

1. History of Type I diabetes mellitus.
2. Pregnancy or breast feeding.
3. Allergy to insulin or insulin products.
4. On-going treatment of steroid-induced hyperglycemia by an endocrinologist and/or general internist.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khanh Vu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vu K, Busaidy N, Cabanillas ME, Konopleva M, Faderl S, Thomas DA, O'Brien S, Broglio K, Ensor J, Escalante C, Andreeff M, Kantarjian H, Lavis V, Yeung SC. A randomized controlled trial of an intensive insulin regimen in patients with hyperglycemic acute lymphoblastic leukemia. Clin Lymphoma Myeloma Leuk. 2012 Oct;12(5):355-62. doi: 10.1016/j.clml.2012.05.004. Epub 2012 Jun 1. PMID 22658895
- See also: University of Texas MD Anderson Cancer Center's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 04/27/2004 through 7/1/2008. All participants recruited at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Fifty-two participants were randomized to a conventional treatment arm or an intensive insulin intervention arm. One participant on the conventional control arm was excluded and did not receive allocated intervention.
Period: Overall Study
Arm/Group | Conventional Care | Intensive Insulin
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Care | Intensive Insulin | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Median (Full Range); unit: years] | 46 [17 to 70] | 57.5 [18 to 85] | 52 [17 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: 1-Year Overall Survival Rate
Description: The overall survival rate defined as percentage of participants in each treatment group who are still alive at 12 months.
Time Frame: 1 year
Population: There were 51 evaluable participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Conventional Care: Control Group - Conventional care using blood sugar management with regular human insulin.
- Intensive Insulin: Intervention Group - Intense blood sugar management with Insulin Aspart + Insulin Glargine
Arm/Group | Conventional Care | Intensive Insulin
Number analyzed (Participants) | 25 | 26
percentage of participants | 80.8 [67 to 97.4] | 63.5 [47 to 85.8]

2. Primary Outcome: Overall Survival
Description: Overall survival (OS) defined as the interval between the date of randomization and the date of death. Calculation of period was from baseline (date of randomization) to the death or last follow-up.
Time Frame: Baseline (date of randomization) to date of death or last follow-up (weekly during treatment then every 2 months post study treatment) up to 6 years
Measure: Median (Full Range); unit: Months
Units Other Than Participants: Deaths
Groups:
- Intervention Group: Intense blood sugar management with Insulin Aspart + Insulin Glargine
Arm/Group | Conventional Care | Intervention Group
Number analyzed (Participants) | 25 | 26
Number analyzed (Deaths) | 8 | 10
Months | 44 [2 to 66] | 62.2 [0.5 to 62.2]

3. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval between the date of complete remission and the date of relapse detection or death. Complete Remission (CR) defined as granulocyte count >1.0 × 10^9/L, platelet count >100 × 10^9/L, no abnormal peripheral blasts, and <5% blasts in normocellular or hypercellular bone marrow.
Time Frame: Date of complete remission to disease progression, assessed for approximately 6 years
Population: There were 51 evaluable participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Conventional Care | Intensive Insulin
Number analyzed (Participants) | 25 | 26
Months | 38.8 [1 to 66] | 24 [1 to 62]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) collection from identification of high blood sugar levels until completion of chemotherapy (about 8 months). Study period was from enrollment beginning on 4/27/2004 and follow up ending on 1/20/2010.
Arm/Group | Conventional Care | Intensive Insulin
Serious Adverse Events (participants affected / at risk) | 9/25 | 10/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Care (N=25) | Intensive Insulin (N=26)
Acute Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Neutropenic Fever (Infections and infestations) | 0 (0) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Death (General disorders) | 8 (8) | 10 (10) — Deaths were due to progressive disease and were not related to the study treatment.

LIMITATIONS AND CAVEATS:
Study terminated early due to futility at the pre-determined interim analysis point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes